CLINICAL TRIAL: NCT02161276
Title: Phase 2 Study of The Optimal Dosage of Tang Ning Tongluo Capsule for Type II Diabetes
Brief Title: Clinical Trials for the Optimal Dosage of Tang Ning Tongluo Capsule
Acronym: TNTL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guizhou Bailing Group Pharmaceutical Co Ltd (Industry)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TNTL-14-01
Record Dates: First submitted 2014-05-21; First posted 2014-06-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Accidental Exposure While Preparing Drug for Administration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TNTL capsule and Placebo (Experimental): 3-4 capsules 3 times a day Used before meals
  Interventions: Drug: TNTL capsule; Drug: Placebo

INTERVENTIONS:
Drug: TNTL capsule — Patients were asked to taken drugs 3 times a day, with each time 3 grains
  Other Names: Tang Ning Tongluo Capsule
Drug: Placebo — Patients were asked to taken drugs 3 times a day, with each time 3 grains

SUMMARY:
Treatment of diabetes mellitus with Traditional Chinese Medicine has a long history.

aim： --establish the optimal dosage of traditional Chinese medicine Tang Ning Tongluo Capsule to treat type II diabetes mellitus.

---Preliminary evaluate the clinical efficacy and safety of Tangning Tongluo Capsule in the treatment of type II diabetes

DETAILED DESCRIPTION:
Preliminary evaluation on the clinical efficacy and safety of Tangning Tongluo Capsule in the treatment of type II diabetes, and provides basis for determining optimal dosage of Tangning Tongluo capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilled diagnostic criteria for type II diabetes and TCM syndrome diagnostic criteria.
2. Age between 18-70 years.
3. The blood sugar meet the following criteria: fasting blood glucose ≥ 7.0mmol/L, ≤ 13 mmol/L and (or) ≥ 2 hour postprandial blood glucose 11.1 mmol/L, ≤ 16 mmol/L; eligible conditions in blood glucose, glycosylated hemoglobin to ≤ 10%.
4. Traditional Chinese medicine symptom score ≥ 4 points.
5. Participated in the experiment voluntarily, and signed the informed consent form.

Exclusion Criteria:

1. Durring the cleaning period, blood sugar dropped to below detection diagnosis value through diet, increasing activity.
2. Secondary diabetes mellitus or nearly a month using insulin; or is the use of insulin sensitizers (thiazolidine two ketones), repaglinide, Bernard Glenn Nai, alpha glucoside enzyme inhibitor (acarbose, voglibose), other traditional Chinese medicine.
3. Within the past 1 months, with diabetic ketoacidosis and other acute metabolic disorders.
4. ALT is 2 times higher than the upper limit of the normal value, Cr is higher than the upper limit of normal persons.
5. Has severe heart, liver, renal, hematopoietic system disease, or other serious diseases and mental disease patients.
6. Pregnant, lactating women and prepare for pregnancy.
7. The allergic constitution and the drug allergy known composition.
8. For nearly a month with severe infection or other emergency state, such as trauma, operation etc..
9. within the past 3 months, participated in the other drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The decline glycosylated hemoglobin A1C and blood glucose level | up to 8 weeks
  Decline in Hemoglobin A1C and blood glucose level

SECONDARY OUTCOMES:
The clinical composite safety evaluation of Tangning Tongluo Capsule in the treatment of type II diabetes participants | 2 months
  Routine check for blood, urine, stool + occult blood, liver function (ALT, AST, AKP, GGT, TBIL), renal function (BuN, Cr), ECG before treatment with 1 times per week.

CONTACTS AND LOCATIONS:
Overall Officials: XY Xin, Dr., Study Director — ICMJE
Locations (1):
- Tianyuan Hospital of Guiyang City, Guiyang, Guizhou, China